CLINICAL TRIAL: NCT00653406
Title: Multiple-dosing Study of Long Acting Injectable of Risperidone in Schizophrenic Patients
Brief Title: A Pharmacokinetic and Safety Study of Risperidone Long Acting Injectable in Schizophrenic Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR003262
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Risperidone; Intramuscular injection; Pharmacokinetics
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Drug: Risperidone long acting injectable

SUMMARY:
The purpose of this study is to explore the pharmacokinetic profile and safety after biweekly (every 2-week) intramuscular (IM) injections (6 injections) of risperidone long acting injectable 25, 37.5, or 50 mg/dose in schizophrenic patients. The efficacy of the study medication will also be assessed.

DETAILED DESCRIPTION:
This is an open-label, multicenter, randomized, 3-arm trial to compare the pharmacokinetic profile and the safety profile between 3 dose groups. There are 2 periods in this study: a 10-week treatment period and an 8-week follow-up period. Patients will receive 6 injections of long acting injectable risperidone at one of the dose levels (25, 37.5 and 50 mg) every 2 weeks according to their randomly assigned treatment. Blood samples will be collected throughout the 10-week treatment and 8-week follow-up period to determine the changes in study drug concentration in the plasma. Safety will be assessed by monitoring of adverse events, subjective symptoms/objective findings, laboratory tests, physical examinations, electrocardiograms, injection site reactions, and the Drug-Induced Extrapyramidal Symptoms Scale (DIEPSS). Efficacy of the study drug will be assessed based on the Positive and Negative Syndrome Scale (PANSS) and the Clinical Global Impression - Severity (CGI-S) and Clinical Global Impression - Change (CGI-C) scales. The patients will receive injections of long acting injectable risperidone (either 25, 37.5, or 50 mg) in their muscle every 2 weeks for 10 weeks for a total of 6 injections.

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients with a DSM-IV diagnosis of schizophrenia
* A Positive and Negative Syndrome Scale (PANSS) total score between 60 (included) and 120 (excluded)
* In- or out-patients (change of institutionalization status during the trial period is allowed).

Exclusion Criteria:

* No DSM-IV diagnosis other than schizophrenia
* No convulsive disorders such as epilepsy
* No neuroleptic malignant syndrome or physical fatigue associated with dehydration, malnutrition
* No present illness or history of diabetes or risks of diabetes such as hyperglycemia and obesity
* No hemorrhagic diathesis.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2002-11; Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
The max and min plasma concentrations, average plasma concentration, and time to reach the max plasma concentration at steady-state (2 weeks after 6th dose). Safety data for all timepoints will be summarized.

SECONDARY OUTCOMES:
The change at Week 12 from the baseline of the total score, positive symptom score, negative symptom score, total psychiatric score and BPRS scores from the PANSS.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.

REFERENCES:
- See also: A pharmacokinetic and safety study of risperidone long acting injectable in schizophrenic patients — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=402&filename=CR003262_CSR.pdf